CLINICAL TRIAL: NCT05241366
Title: Controlled Clinical Trial of Transcranial Magnetic Stimulation Versus Conventional Therapy for the Treatment of Functional Neurological Non-Epileptic Seizure Disorder: A Pilot Study
Brief Title: TMS vs Conventional Therapy for the Treatment of Functional Neurological Non Epileptic Seizure Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez (Other)
Responsible Party: Principal Investigator, Edgar Daniel Crail Melendez, MS, El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16/21
Record Dates: First submitted 2022-01-20; First posted 2022-02-15 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Psychogenic Non-Epileptic Seizure
Keywords: Transcranial Magnetic Stimulation; Selective Serotonin Reuptake Inhibitor; Functional Neurological Disorder
MeSH Terms: conditions — Psychogenic Nonepileptic Seizures; Conversion Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled clinical trial. Non-probabilistic sampling of consecutive cases randomized to each arm of the study. The study will consist of a control group and a study group. The study group will receive a therapeutic scheme with Transcranial Magnetic Stimulation (TMS) + usual pharmacological treatment and the control group will receive an identical scheme with TMS simulated with a sham coil + usual pharmacological treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double masking (Trial Participant/Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Transcranial Magnetic Stimulation + usual treatment with SSRIs (Experimental): Transcranial Magnetic Stimulation + SSRIs The TMS group will be comprised of 10 patients, each subject will receive 12 sessions of low frequency (1 Hz) rTMS over right dorsolateral prefrontal cortex with a total of 1500 each session.
  All patients will continue with the usual treatment established by their treating physician. Those who do not have a previous pharmacological treatment will start a protocol with sertraline, which should be started at a 50 mg/day dosage.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham TMS coil + usual treatment with SSRIs (Sham Comparator): The sham TMS coil group will be comprised of 10 patients, sham TMS stimulation will be performed with the B-65 coil, which has similar sound and scalp contact to those experienced during active stimulation. The duration of treatment will be the same as in the experimental arm.
  All patients will continue with the usual treatment established by their treating physician. Those who do not have a previous pharmacological treatment will start a protocol with sertraline, which should be started at a 50 mg/day dosage.
  Interventions: Device: Sham Transcranial Magnetic Stimulation coil

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — The TMS group will be comprised of 10 patients, each subject will receive 12 sessions of low frequency (1 Hz) rTMS over the right dorsolateral prefrontal cortex with a total of 1500 pulses in each session. Each session will last approximately 30 minutes. There will be one session per day, five sessions per week. The total duration of the treatment will be four weeks.
  All patients will continue with the usual treatment established by their treating physician. Those who do not have a previous pharmacological treatment will start a protocol with sertraline, which should be started at a 50 mg/day dosage.
  Other Names: rTMS
  Arms: Transcranial Magnetic Stimulation + usual treatment with SSRIs
Device: Sham Transcranial Magnetic Stimulation coil — Simulated TMS stimulation will be performed with a Sham TMS coil, which has a sound and scalp contact similar to those experienced during active stimulation. The duration of the treatment will be the same as in the experimental arm.
  All patients will continue with the usual treatment established by their treating physician. Those who do not have a previous pharmacological treatment will start a protocol with sertraline, which should be started at a 50 mg/day dosage.
  Other Names: Sham TMS coil
  Arms: Sham TMS coil + usual treatment with SSRIs

SUMMARY:
The aim of the study is to compare the effect of Transcranial Magnetic Stimulation (TMS) versus treatment with selective serotonin reuptake inhibitors (SSRIs), in patients with diagnosis of Functional Neurological Non Epileptic Seizure Disorder (PNES).

DETAILED DESCRIPTION:
This study consists of a single-blind Randomized Controlled Clinical Trial comprised of 20 patients with diagnosis of Psychogenic Non Epileptic Seizures (PNES), distributed in 2 arms of 10 patients each.

Patients (n=20) will be randomly assigned (using the block randomization method) to one of the groups. Both groups of patients will be receiving their usual medical treatment (SSRIs), one group will receive in addition a therapeutic scheme with active TMS, while the second group will receive the same scheme, but with a sham TMS coil to decrease the bias of placebo effect.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of PNES, based on the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) and the ILAE, confirmed by video recording and/or V-EEG monitoring, and who have a monthly seizure frequency greater than 3.
2. Patients who have a record at the institute with the diagnosis of PNES.
3. Patients with an encephalic MRI.
4. Patients who give their written consent to participate in the protocol.
5. Patients who have not had any changes in the pharmacological treatment in the last 6 weeks.

Exclusion Criteria:

1. Patients who cannot answer the scales and other clinimetric instruments.
2. Patients with a history of previous or current epilepsy.
3. Patients with other major neurological comorbidities (tumor, cerebrovascular event (CVE), cranioencephalic trauma (TBI)).
4. Patients currently taking medications that lower the seizure threshold (Bupropion).
5. Patients with psychiatric comorbidities such as psychosis/bipolar disorder/substance abuse.
6. Patients with certain implanted metallic devices (pacemakers).
7. Pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
PNES count (1/4) | Baseline PNES count (Starting 1 month before TMS treatment)
  Participants in both groups will registered in a specific chart, daily psychogenic non-epileptic seizure activity.
PNES count (2/4) | Change from Baseline PNES count (immediately after the session 12th -last session-)
  Participants in both groups will registered in a specific chart, daily psychogenic non-epileptic seizure activity.
PNES count (3/4) | Change from Baseline PNES count at month 1 post treatment
  Participants in both groups will registered in a specific chart, daily psychogenic non-epileptic seizure activity.
PNES count (4/4) | Change from Baseline PNES count at month 2 post treatment
  Participants in both groups will registered in a specific chart, daily psychogenic non-epileptic seizure activity.

SECONDARY OUTCOMES:
Psychometric self-assessment scales (BDI-II) 1/4 | Baseline score (1 month before TMS treatment)
  1.0) Mood: Beck Depression Inventory-II (BDI-II)
  Minimum score: 0
  Maximum score: 63
  1-10: These ups and downs are considered normal
  11-16: Mild mood disturbance
  17-20: Borderline clinical depression
  21-30: Moderate depression
  31-40: Severe depression
  over 40: Extreme depression
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (BDI-II) 2/4 | Change from Baseline score (immediately after the 12th session -last session-)
  1.1) Mood: Beck Depression Inventory-II (BDI-II)
  Minimum score: 0
  Maximum score: 63
  1-10: These ups and downs are considered normal
  11-16: Mild mood disturbance
  17-20: Borderline clinical depression
  21-30: Moderate depression
  31-40: Severe depression
  over 40: Extreme depression
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (BDI-II) 3/4 | Change from Baseline score at month 1 post treatment
  1.2) Mood: Beck Depression Inventory-II (BDI-II)
  Minimum score: 0
  Maximum score: 63
  1-10: These ups and downs are considered normal
  11-16: Mild mood disturbance
  17-20: Borderline clinical depression
  21-30: Moderate depression
  31-40: Severe depression
  over 40: Extreme depression
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (BDI-II) 4/4 | Change from Baseline score at month 2 post treatment
  1.3) Mood: Beck Depression Inventory-II (BDI-II)
  Minimum score: 0
  Maximum score: 63
  1-10: These ups and downs are considered normal
  11-16: Mild mood disturbance
  17-20: Borderline clinical depression
  21-30: Moderate depression
  31-40: Severe depression
  over 40: Extreme depression
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (DES) 1/4 | Baseline score (1 month before TMS treatment)
  2.0) Dissociation : Dissociative Experience Scale (DES).
  Minimum score: 0
  Maximum score: 100
  High levels of dissociation are indicated by scores of 30 or more, scores under 30 indicate low levels.
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (DES) 2/4 | Change from Baseline score (immediately after the 12th session -last session-)
  2.1) Dissociation : Dissociative Experience Scale (DES).
  Minimum score: 0
  Maximum score: 100
  High levels of dissociation are indicated by scores of 30 or more, scores under 30 indicate low levels.
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (DES) 3/4 | Change from Baseline score at month 1 post treatment
  2.2) Dissociation : Dissociative Experience Scale (DES).
  Minimum score: 0
  Maximum score: 100
  High levels of dissociation are indicated by scores of 30 or more, scores under 30 indicate low levels.
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (DES) 4/4 | Change from Baseline score at month 2 post treatment
  2.3) Dissociation : Dissociative Experience Scale (DES).
  Minimum score: 0
  Maximum score: 100
  High levels of dissociation are indicated by scores of 30 or more, scores under 30 indicate low levels.
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (PTSD) 1/4 | Baseline score (1 month before TMS treatment)
  3.0) PTSD/Trauma/Resilience: PTSD Symptom Severity Scale.
  Minimum score: 0
  Maximum score: 80
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (PTSD) 2/4 | Change from Baseline score (immediately after the 12th session -last session-)
  3.1) PTSD/Trauma/Resilience: PTSD Symptom Severity Scale.
  Minimum score: 0
  Maximum score: 80
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (PTSD) 3/4 | Change from Baseline score at month 1 post treatment
  3.2) PTSD/Trauma/Resilience: PTSD Symptom Severity Scale.
  Minimum score: 0
  Maximum score: 80
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (PTSD) 4/4 | Change from Baseline score at month 2 post treatment
  3.3) PTSD/Trauma/Resilience: PTSD Symptom Severity Scale.
  Minimum score: 0
  Maximum score: 80
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (MoCA) 1/4 | Baseline score (1 month before TMS treatment)
  4.0) Education and Cognition: Montreal Cognitive Assessment (MoCA).
  Minimum score: 0
  Maximum score: 30
  Normal score: 26-30
  Probable Neurocognitive Dissorder: 0-25
  *Higher scores mean a better outcome.
Psychometric self-assessment scales (MoCA) 2/4 | Change from Baseline score (immediately after the 12th session -last session-)
  4.1) Education and Cognition: Montreal Cognitive Assessment (MoCA).
  Minimum score: 0
  Maximum score: 30
  Normal score: 26-30
  Probable Neurocognitive Dissorder: 0-25
  *Higher scores mean a better outcome.
Psychometric self-assessment scales (MoCA) 3/4 | Change from Baseline score at month 1 post treatment
  4.2) Education and Cognition: Montreal Cognitive Assessment (MoCA).
  Minimum score: 0
  Maximum score: 30
  Normal score: 26-30
  Probable Neurocognitive Dissorder: 0-25
  *Higher scores mean a better outcome.
Psychometric self-assessment scales (MoCA) 4/4 | Change from Baseline score at month 2 post treatment
  4.3) Education and Cognition: Montreal Cognitive Assessment (MoCA).
  Minimum score: 0
  Maximum score: 30
  Normal score: 26-30
  Probable Neurocognitive Dissorder: 0-25
  *Higher scores mean a better outcome.
Psychometric self-assessment scales (WHOQOL-BREF) 1/4 | Baseline score (1 month before TMS treatment)
  5.0) Quality of life: WHOQOL-BREF (World Health Organization Quality of Life-BREF).
  Minimum score: 0
  Maximum score: 100
  *Higher scores mean a better outcome.
Psychometric self-assessment scales (WHOQOL-BREF) 2/4 | Change from Baseline score (immediately after the 12th session -last session-)
  5.1) Quality of life: WHOQOL-BREF (World Health Organization Quality of Life-BREF).
  Minimum score: 0
  Maximum score: 100
  *Higher scores mean a better outcome.
Psychometric self-assessment scales (WHOQOL-BREF) 3/4 | Change from Baseline score at month 1 post treatment
  5.2) Quality of life: WHOQOL-BREF (World Health Organization Quality of Life-BREF).
  Minimum score: 0
  Maximum score: 100
  *Higher scores mean a better outcome.
Psychometric self-assessment scales (WHOQOL-BREF) 4/4 | Change from Baseline score at month 2 post treatment
  5.3) Quality of life: WHOQOL-BREF (World Health Organization Quality of Life-BREF).
  Minimum score: 0
  Maximum score: 100
  *Higher scores mean a better outcome.
Psychometric self-assessment scales (King's) 1/4 | Baseline score (1 month before TMS treatment)
  6.0) King's Internalized Stigma Scale.
  Minimum score: 0
  Maximum score: 112
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (King's) 2/4 | Change from Baseline score (immediately after the 12th session -last session-)
  6.1) King's Internalized Stigma Scale.
  Minimum score: 0
  Maximum score: 112
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (King's) 3/4 | Change from Baseline score at month 1 post treatment
  6.2) King's Internalized Stigma Scale.
  Minimum score: 0
  Maximum score: 112
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (King's) 4/4 | Change from Baseline score at month 2 post treatment
  6.3) King's Internalized Stigma Scale.
  Minimum score: 0
  Maximum score: 112
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (OCI-R) 1/4 | Baseline score (1 month before TMS treatment)
  7.0) Obsessions/compulsions: The Obsessive-Compulsive Inventory Short Version (OCI-R)
  Minimum score: 0
  Maximum score: 72
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (OCI-R) 2/4 | Change from Baseline score (immediately after the 12th session -last session-)
  7.1) Obsessions/compulsions: The Obsessive-Compulsive Inventory Short Version (OCI-R)
  Minimum score: 0
  Maximum score: 72
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (OCI-R) 3/4 | Change from Baseline score at month 1 post treatment
  7.2) Obsessions/compulsions: The Obsessive-Compulsive Inventory Short Version (OCI-R)
  Minimum score: 0
  Maximum score: 72
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (OCI-R) 4/4 | Change from Baseline score at month 2 post treatment
  7.3) Obsessions/compulsions: The Obsessive-Compulsive Inventory Short Version (OCI-R)
  Minimum score: 0
  Maximum score: 72
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (BAI) 1/4 | Baseline score (1 month before TMS treatment)
  8.0) Beck Anxiety Inventory (BAI).
  Minimum score: 0
  Maximum score: 63
  Minimal: 0 - 7
  Mild: 8 - 15
  Moderate: 16 - 25
  Severe: 26 - 63
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (BAI) 2/4 | Change from Baseline score (immediately after the 12th session -last session-)
  8.1) Beck Anxiety Inventory (BAI).
  Minimum score: 0
  Maximum score: 63
  Minimal: 0 - 7
  Mild: 8 - 15
  Moderate: 16 - 25
  Severe: 26 - 63
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (BAI) 3/4 | Change from Baseline score at month 1 post treatment
  8.2) Beck Anxiety Inventory (BAI).
  Minimum score: 0
  Maximum score: 63
  Minimal: 0 - 7
  Mild: 8 - 15
  Moderate: 16 - 25
  Severe: 26 - 63
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (BAI) 4/4 | Change from Baseline score at month 2 post treatment
  8.3) Beck Anxiety Inventory (BAI).
  Minimum score: 0
  Maximum score: 63
  Minimal: 0 - 7
  Mild: 8 - 15
  Moderate: 16 - 25
  Severe: 26 - 63
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (HADS) 1/4 | Baseline score (1 month before TMS treatment)
  9.0) Anxiety: Hospital Anxiety and Depression Scale (HADS).
  Depression (D):
  Minimum score: 0
  Maximum score: 21
  Anxiety (A):
  Minimum score: 0
  Maximum score: 21
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (HADS) 2/4 | Change from Baseline score (immediately after the 12th session -last session-)
  9.1) Anxiety: Hospital Anxiety and Depression Scale (HADS).
  Depression (D):
  Minimum score: 0
  Maximum score: 21
  Anxiety (A):
  Minimum score: 0
  Maximum score: 21
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (HADS) 3/4 | Change from Baseline score at month 1 post treatment
  9.2) Anxiety: Hospital Anxiety and Depression Scale (HADS).
  Depression (D):
  Minimum score: 0
  Maximum score: 21
  Anxiety (A):
  Minimum score: 0
  Maximum score: 21
  *Higher scores mean a worse outcome.
Psychometric self-assessment scales (HADS) 4/4 | Change from Baseline score at month 2 post treatment
  9.3) Anxiety: Hospital Anxiety and Depression Scale (HADS).
  Depression (D):
  Minimum score: 0
  Maximum score: 21
  Anxiety (A):
  Minimum score: 0
  Maximum score: 21
  *Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Édgar Daniel Crail Meléndez, MD, Principal Investigator — Instituto Nacional de Neurología y Neurocirugía Manuel Velasco Suárez
Locations (1):
- Instituto Nacional de Neurologia Y Neurocirugia Mvs, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agarwal R, Garg S, Tikka SK, Khatri S, Goel D. Successful use of theta burst stimulation (TBS) for treating psychogenic non epileptic seizures (PNES) in a pregnant woman. Asian J Psychiatr. 2019 Jun;43:121-122. doi: 10.1016/j.ajp.2019.05.013. Epub 2019 May 8. No abstract available. PMID 31125954
- [Background] LaFrance, W., & Blumer, D. (2018). Pharmacological Treatments for Psychogenic Nonepileptic Seizures. University of Warwick. Retrieved from: https://www.cambridge.org/core.
- [Background] LaFrance WC Jr, Keitner GI, Papandonatos GD, Blum AS, Machan JT, Ryan CE, Miller IW. Pilot pharmacologic randomized controlled trial for psychogenic nonepileptic seizures. Neurology. 2010 Sep 28;75(13):1166-73. doi: 10.1212/WNL.0b013e3181f4d5a9. Epub 2010 Aug 25. PMID 20739647
- [Background] Varia I, Logue E, O'connor C, Newby K, Wagner HR, Davenport C, Rathey K, Krishnan KR. Randomized trial of sertraline in patients with unexplained chest pain of noncardiac origin. Am Heart J. 2000 Sep;140(3):367-72. doi: 10.1067/mhj.2000.108514. PMID 10966532
- [Background] Peterson, K., et al. (2017). Transcranial Magnetic Stimulation in the treatment of non-epileptic seizures: A Case Series. Max Rady College of Medicine. University of Manitoba.
- [Background] Peterson KT, Kosior R, Meek BP, Ng M, Perez DL, Modirrousta M. Right Temporoparietal Junction Transcranial Magnetic Stimulation in the Treatment of Psychogenic Nonepileptic Seizures: A Case Series. Psychosomatics. 2018 Nov;59(6):601-606. doi: 10.1016/j.psym.2018.03.001. Epub 2018 Mar 7. PMID 29628295
- [Background] Benbadis SR, Allen Hauser W. An estimate of the prevalence of psychogenic non-epileptic seizures. Seizure. 2000 Jun;9(4):280-1. doi: 10.1053/seiz.2000.0409. PMID 10880289
- [Background] Duncan R, Razvi S, Mulhern S. Newly presenting psychogenic nonepileptic seizures: incidence, population characteristics, and early outcome from a prospective audit of a first seizure clinic. Epilepsy Behav. 2011 Feb;20(2):308-11. doi: 10.1016/j.yebeh.2010.10.022. Epub 2010 Dec 30. PMID 21195031
- [Background] Kanemoto K, LaFrance WC Jr, Duncan R, Gigineishvili D, Park SP, Tadokoro Y, Ikeda H, Paul R, Zhou D, Taniguchi G, Kerr M, Oshima T, Jin K, Reuber M. PNES around the world: Where we are now and how we can close the diagnosis and treatment gaps-an ILAE PNES Task Force report. Epilepsia Open. 2017 Jun 23;2(3):307-316. doi: 10.1002/epi4.12060. eCollection 2017 Sep. PMID 29588959
- [Background] Pollak TA, Nicholson TR, Edwards MJ, David AS. A systematic review of transcranial magnetic stimulation in the treatment of functional (conversion) neurological symptoms. J Neurol Neurosurg Psychiatry. 2014 Feb;85(2):191-7. doi: 10.1136/jnnp-2012-304181. Epub 2013 Jan 8. PMID 23303960
- [Background] Dafotakis M, Ameli M, Vitinius F, Weber R, Albus C, Fink GR, Nowak DA. [Transcranial magnetic stimulation for psychogenic tremor - a pilot study]. Fortschr Neurol Psychiatr. 2011 Apr;79(4):226-33. doi: 10.1055/s-0029-1246094. Epub 2011 Apr 8. German. PMID 21480152
- [Background] van der Kruijs SJ, Bodde NM, Vaessen MJ, Lazeron RH, Vonck K, Boon P, Hofman PA, Backes WH, Aldenkamp AP, Jansen JF. Functional connectivity of dissociation in patients with psychogenic non-epileptic seizures. J Neurol Neurosurg Psychiatry. 2012 Mar;83(3):239-47. doi: 10.1136/jnnp-2011-300776. Epub 2011 Nov 5. PMID 22056967
- [Background] van der Kruijs SJ, Jagannathan SR, Bodde NM, Besseling RM, Lazeron RH, Vonck KE, Boon PA, Cluitmans PJ, Hofman PA, Backes WH, Aldenkamp AP, Jansen JF. Resting-state networks and dissociation in psychogenic non-epileptic seizures. J Psychiatr Res. 2014 Jul;54:126-33. doi: 10.1016/j.jpsychires.2014.03.010. Epub 2014 Mar 21. PMID 24703187
- [Background] Parain D, Chastan N. Large-field repetitive transcranial magnetic stimulation with circular coil in the treatment of functional neurological symptoms. Neurophysiol Clin. 2014 Oct;44(4):425-31. doi: 10.1016/j.neucli.2014.04.004. Epub 2014 May 15. PMID 25306083
- [Background] Nightscales R, McCartney L, Auvrez C, Tao G, Barnard S, Malpas CB, Perucca P, McIntosh A, Chen Z, Sivathamboo S, Ignatiadis S, Jones S, Adams S, Cook MJ, Kwan P, Velakoulis D, D'Souza W, Berkovic SF, O'Brien TJ. Mortality in patients with psychogenic nonepileptic seizures. Neurology. 2020 Aug 11;95(6):e643-e652. doi: 10.1212/WNL.0000000000009855. Epub 2020 Jul 20. PMID 32690794